CLINICAL TRIAL: NCT06381115
Title: An App-Based, Precision Medicine Approach to Optimize Long-Term CPAP Adherence and Quality of Life
Brief Title: App-Based Optimization of Long-Term CPAP Adherence and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (ASU) (Unknown)
Responsible Party: Principal Investigator, Timothy Morgenthaler, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-006685
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SleepWell24 Smart Application (Experimental): This group will consists of participates who will be on study for 8 weeks using the Sleepwell24 application. Once 20 people are enrolled on the 8 week cohort, a 6 month cohort will open up for 20 different participants.
  Interventions: Behavioral: SleepWell24 Application

INTERVENTIONS:
Behavioral: SleepWell24 Application — The SleepWell24 application will use connections with a Shelly smart plug and a Fitbit Charge 4 along with weekly questionnaires to monitor CPAP usage.

SUMMARY:
The purpose of this study is to optimize the time of CPAP usage to at least 6 hours a night for 6 nights per week for people who have OSA with the help of a smartphone application called SmartWell24. This application aims to target CPAP adherence.

ELIGIBILITY:
Inclusion Criteria:

* In both trials of Aim 2, twenty adults (≥18 years) per trial will be recruited who are newly diagnosed with OSA and speak English.
* In both trials, we will purposely recruit samples balanced by biological sex and OSA severity (apnea hypopnea index: 5-14 vs. ≥ 15).
* Inclusion Criteria are the same for both Aim 2 trials; Adult patients from MCCSM sites who:

  * Are diagnosed with OSA based on clinical diagnostic testing via laboratory or home-based sleep study;
  * Own and have the functional and cognitive ability to use an Apple (iOS9 or higher) or Android (4.2 or higher) smartphone with minimal to no assistance;
  * Are prescribed continuous or auto-titrated CPAP;
  * Agree to using a smartphone application and wearable wrist sensor; and
  * Speak and read English.

Exclusion Criteria:

* Unwilling to complete study measures and engage with SleepWell24;
* Refuse to not use the Fitbit application during the study trial;
* Have any conditions that would impede full participation (e.g., communication or cognitive impairments that limit ability to read and/or follow directions, other acute or severe health, cognitive, or psychological conditions);
* Currently participating in other lifestyle programs (e.g. active, formal weight loss program or research study; smoking cessation program, etc.);
* Decide to use a different PAP device than ResMed Airsense 10;
* Prescribed high-dose benzodiazepines (equivalent to > 1 mg lorazapam/night);
* Daily opioid medication use at night;'
* Unwilling to discontinue use of any current wearable sensor for the duration of the trial;
* Previous documented history of treatment/referral for claustrophobia;
* Previous CPAP use;
* Currently engaging in shiftwork defined as night shift or rotating day and night shifts; and
* Currently pregnant, trying to conceive, or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
CPAP Adoption | approximately 6 months
  The Shelly smart plug will be used to monitor the amount of CPAP time usage by the amount of wattage recorded.
Change in Quality of Life | baseline, weekly assessments for approximately 6 months
  As measured by weekly survey asking participants to rate their health based on excellent, very good, good, fair, and poor.

SECONDARY OUTCOMES:
Change in sleep time | baseline, weekly assessments for approximately 6 months
  As measured by the Fitbit Charge 4 sensor, reported in hours
Change in physical activity | baseline, weekly assessments for approximately 6 months
  As measured by the Fitbit Charge 4 sensor step count, reported as number of steps taken daily
Change in sedentary time | baseline, weekly assessments for approximately 6 months
  As measured by the Fitbit Charge 4 sensor, reported in hours

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morgenthaler, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials